CLINICAL TRIAL: NCT04532697
Title: Efficacy of Uncaria Rhynchophylla (Gou-Teng) for Patients With Mild Cognitive Impairment: A Pilot Randomized Controlled Trial Using White Matter Hyperintensities Estimated by ARIA as Outcome
Brief Title: Use of Gou-Teng to Treat Patients With Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-Gou Teng study
Record Dates: First submitted 2020-07-22; First posted 2020-08-31 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Mild Cognitive Impairment; White Matter Hyperintensity
Keywords: Gou-Teng; Mild Cognitive Impairment; White Matter Hyperintensities; ARIA
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Uncaria rhynchophylla

STUDY DESIGN:
Intervention Model Description: All patients will recruited in parallel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All the participants, outcome assessors and the investigator are all masked, only the staff preparing the study product know the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese Medicine (Active Comparator): Uncaria Rhynchophylla (Gou-Teng)
  Interventions: Other: Uncaria Rhynchophylla (Gou-Teng)
- Placebo treatment (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Uncaria Rhynchophylla (Gou-Teng) — Uncaria Rhynchophylla (Gou-Teng) is a kind of Chinese Medicine. All eligible subjects will be randomly assigned to receive a treatment of either Uncaria Rhynchophylla or placebo for 16 weeks followed by 8 weeks observation. The patient will be asked to take 1.2 g of the granule in the morning and another 1.2 g in the evening.
  Arms: Chinese Medicine
Other: Placebo — All eligible subjects will be randomly assigned to receive a treatment of either Uncaria Rhynchophylla or placebo for 16 weeks followed by 8 weeks observation. The patient will be asked to take 1.2 g of the granule in the morning and another 1.2 g in the evening.
  Arms: Placebo treatment

SUMMARY:
Mild cognitive impairment (MCI) is a pre-dementia condition commonly occurs in elderly people. As Hong Kong has become an aged society, the prevalence of dementia and MCI in Hong Kong has increased substantially in recent decades. To date, no effective pharmacological therapies are available for MCI, and there exists a need for exploring complementary treatment for this age-related condition. Preclinical studies have identified Uncaria rhynchophylla (Gouteng in Chinese) to have promising neuroprotective effect in Alzheimer's disease experimental models.

Objective: To assess the effectiveness and the safety of oral administration of Uncaria rhynchophylla for MCI in older people in Hong Kong.

Study design: This is a double-blinded, randomized, placebo controlled pilot study. 56 patients with MCI will be randomized into two groups i.e. Uncaria rhynchophylla and placebo groups. All subjects will receive treatment twice a day for a consecutive 16 weeks.

DETAILED DESCRIPTION:
It is hypothesized that U. rhynchophylla may have good therapeutic efficacy for the treatment of MCI. However, up to now, there exists no clinical data to support the use of U.rhynchophylla for MCI. To evaluate the efficacy of U. rhynchophylla for MCI, the investigator will use a fully automatic retinal image analysis (ARIA) method to estimate the WMH and use this as one of the outcome measures.

The aim of this pilot study is to evaluate the effectiveness and safety of a Chinese herbal preparation U. rhynchophylla for subjects with mild cognitive impairment. It is hypothesized that treatment with U. rhynchophylla is able to significantly improve the cognitive function of subjects with MCI and reduce the white matter hyperintensities (WMH) in the brain of these subjects.

All eligible subjects will be randomly assigned to receive a treatment of either Uncaria rhynchophylla or placebo for 16 weeks followed by 8 weeks observation. All subjects, both of the intervention and control group, will receive standard routine care from the conventional healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female individuals aged 65 years or over at their last birthday
* Montreal Cognitive Assessment (Hong Kong version) (HK-MoCA) age/education matched percentile (score), with the cut off score of ≤16th percentile
* Understand the questionnaires used in the study
* Agreement to give informed consent

Exclusion Criteria:

* Known dementia including Alzheimer's disease
* Current drug use for the treatment of MCI or dementia
* Patient Health Questionnaire-9 (PHQ-9) score 15 or more
* Known psychiatric diseases such as depressive episode, bipolar disorder, obsessive-compulsive disorder and schizophrenia;
* Known history of seizures;
* Known history of stroke associated with permanent disability;
* Known history of liver and renal impairment;
* Known history of allergy to Chinese herbal medicine;
* Concomitant use of warfarin or any anti-coagulants
* Current history of hazardous or harmful alcohol consumption;
* Current medical history that prevented participation in the study tasks such as sensory impairment and advanced cancer;
* Current use of any kind of herbal medicine for the prevention and treatment of dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
HK-MoCA | 16 weeks
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. Scoring of HK MoCA ranges from 0 to 30 points. 3 cutoff percentile will be used: 2nd, 7th, and 16th percentile. The cut-off percentile at 16th above is considered normal and it shows worse with the decreasing percentile.

SECONDARY OUTCOMES:
Automatic Retinal Image Analysis (ARIA) | 16 weeks
  White Matter Hyperintensities (WMH) is closely associated with multiple brain functions. It is an objective surrogate marker for MCI/dementia. The severity of WMH changes can be estimated by taking the fundus retinal image and put to the ARIA algorithm, the scale ranges from 0 to 3, increasing score means increasing severity.
HK-MoCA | 24 weeks
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. Scoring of HK MoCA ranges from 0 to 30 points. 3 cutoff percentile will be used: 2nd, 7th, and 16th percentile. The cut-off percentile at 16th above is considered normal and it shows worse with the decreasing percentile.
Automatic Retinal Image Analysis (ARIA) | 24 weeks
  White Matter Hyperintensities (WMH) is closely associated with multiple brain functions. It is an objective surrogate marker for MCI/dementia. The severity of WMH changes can be estimated by taking the fundus retinal image and put to the ARIA algorithm, the scale ranges from 0 to 3, increasing score means increasing severity.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No